CLINICAL TRIAL: NCT03746873
Title: A Web-based Self-management Intervention to Increase Level of Physical Activity and Decrease Use of Health Care for People With COPD, in Primary Care: A Protocol for a Randomized Controlled Clinical Trial
Brief Title: Increase Level of Physical Activity and Decrease Use of Health Care for People With COPD
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KOLwebben1
Record Dates: First submitted 2018-11-15; First posted 2018-11-20 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Health promotion tool; Self management; Evidence based care; Implementation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD Web (Experimental): Participants randomised to experimental group will be introduced to the COPD Web by a letter containing written information. All participants will receive a pedometer and written information about the importance of physical activity.
  Interventions: Behavioral: COPD Web
- Control (No Intervention): Other than receiving a pedometer and written information about the importance of physical activity the patients in the control group will not receive any intervention.

INTERVENTIONS:
Behavioral: COPD Web — The COPD Web will be introduced to the participant randomized to intervention by a letter containing a code to get access to the web site and how to create an account and login. At the web site there will be an instruction movie showing/ discussing specific content on the COPD Web. The web site will be self-managed. To secure that there is no technical or user problems participants will be contacted by a researcher the first week of intervention.
  Participants will receive "push notifications" (email) with targeted information containing links to the COPD Web and reminder to register the number of steps walked during that week. The push notifications will come every week (week 1-12), every other week (week 12 to 24) and every fourth week (week 24-52).
  Arms: COPD Web

SUMMARY:
This study evaluates the effects of the COPD Web (KOLwebben), an interactive web-based tool directed towards people with chronic obstructive pulmonary disease (COPD). The COPD Web include tools that improve health literacy with a specific focus on 1) increased physical activity and 2) use of appropriate self-management strategies. This randomized clinical trial aims to generate evidence on the effect and usability of the COPD Web in a properly powered cohort of patients in primary care context.

DETAILED DESCRIPTION:
COPD is a chronic and disabling disease with substantial morbidity and mortality. The disease is one of the top 5 leading causes of death worldwide and the high prevalence places a considerable burden on the health care system. The symptom burden of the disease; dyspnea, fatigue, impaired functional performance, decreased level of physical activity and quality of life in patients with COPD are not only a consequence of the underlying condition, but depend also on the patients' adaptation to the symptoms and their ability to manage their disabling disease.

Self-management strategies, including strategies to promote self-efficacy through increasing the patients' knowledge, skills and their confidence in successfully managing their chronic disease is therefore an important part of COPD management. Even though education and promotion of self-management strategies for patients with COPD could be performed independently using a case manager, it is often promoted through pulmonary rehabilitation. In this context self-management means supporting individuals in gaining personal care and health behavioral skills, and develops confidence in applying these skills in everyday life. Pulmonary rehabilitation has been shown to be cost effective and is recommended as treatment for people with mild to very severe COPD since regular physical activity reduces hospital admissions and mortality in COPD. Support for self-management and education is often promoted by an asthma/COPD-nurse through pulmonary rehabilitation. However, in Sweden only a limited proportion of patients with COPD get access to such services which is related to both structural as well as individual barriers. With regard to the former, both limited access to pulmonary rehabilitation as well as to relevant health professionals have recently been reported in Swedish primary care settings. Individual barriers for participation in pulmonary rehabilitation programs found among patients with COPD are lack in knowledge and insight in their diagnosis, transportation and changing health.

Consequently there is an urgent need to find new strategies to facilitate the provision of self-management support to patients with COPD. Electronic health (eHealth) solutions are a promising way of delivering health service, and has previously been used as an alternative way of delivering pulmonary rehabilitation to patients with COPD. However, even though eHealth solutions have been suggested to have the potential to deliver support for self-management in patients with COPD, effects are inconsistent and further research is warranted. Therefore, to further address this question, the research group have developed the COPD Web, a web-based tool aimed at facilitating support for self-management through increasing the patients' knowledge and skills. The COPD Web has been co-created together with health professionals, patients with COPD, their relatives and experts in pulmonary rehabilitation. The COPD Web includes, in addition to texts, pictures and films (e.g., how to perform exercise training, breathing techniques etc.) also interactive components, such as a tool for registration of steps per day with automatized feedback. In a pilot study on 83 patients the investigators found promising results showing increased self-reported level of physical activity that is of great interest since level of physical activity is the strongest predictor of mortality in COPD. However, the pilot study fell short in design, i.e the intervention was not randomized, and there were a lack of power and objective measurements. Still, studies evaluating whether an objective web-based tool as the COPD Web could be used to promote self-management strategies in order to support e.g. increased physical activity in patients with COPD are contradictory and so far no study has been performed in a Swedish context.

The design will be a randomized controlled clinical trial with a baseline assessment and 3- and 12-months follow up regarding effects on physical activity, health related quality of life, COPD related symptoms and health economics as a consequence of the use of the COPD Web. In addition will the investigators identify enablers and barriers for the use of an web-based solution like the COPD Web in order to change behavior. All persons with COPD who visits included primary care centres in Sweden, until a total of 144 participants are included will constitute the sample in the intervention (COPD Web) and control group.

ELIGIBILITY:
Inclusion Criteria:

* All persons with a diagnosis of COPD (ICD-10:J44:9) who visit included primary care units due to their COPD.
* Needs to understand and read Swedish.
* Needs to have a smartphone, tablet or computer with access to internet.
* In case of exacerbation, the participant has to wait at least 6 weeks after initiated pharmacological treatment, before being eligible in the study.

Exclusion Criteria:

* Not COPD
* Dementia or other psychiatric condition that can prevent understanding of the intervention.
* Serious comorbidity that can be considered as the contributing factor for limitation in physical activity.
* Has an account on the COPD Web.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Change in level of objectively measured physical activity | 7 Days at baseline, 7 days at 3- and 12- months after baseline
  Level of physical activity will be objectively measured with an activity monitor, the DynaPort MiniMod. The activity monitor data collected during 7 Days at baseline and 7 Days 3- and 12- months after baseline will be used to assess change in level of physical activity.

SECONDARY OUTCOMES:
Change in level of subjectively assessed physical activity | 7 Days at baseline, 7 days at 3- and 12- months after baseline
  Level of physical activity will be subjectively assessed with Socialstyrelsens indicator questions on physical activity.
Change in subjectively assessed dyspnea severity | 7 Days at baseline, 7 days at 3- and 12- months after baseline
  Dyspnea severity will be assessed using the modified Medical Research Council dyspnea scale (mMRC)
Change in subjectively assessed COPD-related symptoms | 7 Days at baseline, 7 days at 3- and 12- months after baseline
  Change in COPD-related symptoms will be assessed using the COPD assessment test (CAT).
Change in subjectively assessed health related quality of life | 7 Days at baseline, 7 days at 3- and 12- months after baseline
  Change in health related quality of life will be assessed using the Chronic Respiratory Questionnaire, self-administered (CRQ-SA)
Change in health economics using subjectively assessed EQ-5D in combination with self-reported health care contacts | 7 Days at baseline, 7 days at 3- and 12- months after baseline
  Evaluation of health economics will be done using EQ-5D in combination with the number of COPD-related health care contacts that will be self-reported.

OTHER OUTCOMES:
Enablers and barriers for the use of COPD Web in order to change behavior. | 3 months after baseline
  Semi structured interviews and content analysis will be performed in a subgroup of patients randomized to intervention to identify enablers and barriers for the use of an eHealth solution like COPD Web in order to change behavior. The patients will receive a question to take part in an interview at the 3 month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Wadell, PhD, Principal Investigator — Umeå University; Tobias Stenlund, PhD, Study Director — Umeå University; André Nyberg, PhD, Study Director — Umeå University; Sara Lundell, MSc, Study Director — Umeå University
Locations (1):
- Umeå university, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stenlund T, Nyberg A, Lundell S, Wadell K. Web-based support for self-management strategies versus usual care for people with COPD in primary healthcare: a protocol for a randomised, 12-month, parallel-group pragmatic trial. BMJ Open. 2019 Oct 7;9(10):e030788. doi: 10.1136/bmjopen-2019-030788. PMID 31594889
- See also: The COPDwebb is the site that participants in the intervention group will get access to. The site is locked with password during the study. People otside the study may still use the site with password kol1. — http://www.kolwebben.se/

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT03746873/SAP_000.pdf